CLINICAL TRIAL: NCT03300349
Title: Interhospital Variability in Programmes to Prevent Axillary Lymphadenectomy Sequels in Breast Cancer Patients.
Status: Completed | Type: Observational
Sponsor: Violeta Pajero Otero (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); University of Castilla-La Mancha (Other); Puerta de Hierro University Hospital (Other); Complejo Hospitalario Universitario de Cartagena (Unknown)
Responsible Party: Sponsor-Investigator, Violeta Pajero Otero, Physiotherapist at the Mammary Pathology Unit, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: InveCuidRh001
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer Lymphedema; Shoulder Injury
Keywords: Breast cancer; Breast cancer-related lymphedema; Shoulder injury; Prevention; Educational activity; Physiotherapy
MeSH Terms: conditions — Breast Cancer Lymphedema; Shoulder Injuries; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- axillary lymphadenectomy sequels: Patients who have suffered from axillary lymphadenectomy due to breast cancer between 2014 and 2016 and who have developed breast cancer-related lymphedema and/or shoulder disability who fulfill or not a preventive programme
  Interventions: Other: Fulfillment of a preventive programme; Other: No fulfillment of a preventive programme
- No axillary lymphadenectomy sequels: Patients who have suffered from axillary lymphadenectomy due to breast cancer between 2014 and 2016 and who have not develped breast cancer-related lymphedema and/or shoulder disability who fulfill or not a preventive programme.
  Interventions: Other: Fulfillment of a preventive programme; Other: No fulfillment of a preventive programme
- Fulfillment of a preventive programme: Patients who fulfil a preventive programme for axillary lymphadenectomy sequels
- No fulfillment of a preventive programme: Patients who do not fulfil a preventive programme for axillary lymphadenectomy sequels

INTERVENTIONS:
Other: Fulfillment of a preventive programme — Information about risk factors for breast cancer-related lymphedema and home-based exercise programme for shoulder
  Groups: No axillary lymphadenectomy sequels; axillary lymphadenectomy sequels
Other: No fulfillment of a preventive programme — No fulfillment of the preventive programme: Information about risk factors for breast cancer-related lymphedema and home-based exercise programme for shoulder
  Groups: No axillary lymphadenectomy sequels; axillary lymphadenectomy sequels

SUMMARY:
This study aims to determine the effectiveness of the different programmes of four Spanish hospitals about prevention of axillary lymphadenectomy sequels in breast cancer patients.

DETAILED DESCRIPTION:
This study aims to describe the different programs for the prevention of sequels of axillary lymphadenectomy in patients with breast cancer in four Spanish hospitals, to determine the degree of compliance of these programs and to register the frecuency of lymphedema and limitation of mobility of the upper limb in breast cancer patients undergoing axillary lymphadenectomy between 2014 and 2016 in the four hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from axillary lymphadenectomy due to breast cancer treatment between 1 january 2014 until 31 december 2016.

Exclusion Criteria:

* Lymphedema prior to surgery in any of the upper limbs or any malformation or injury that prevents comparison of both upper limb volumes.
* Cognitive impairment or intellectual disability that would prevent understanding the instructions of the study, as well as the purpose of the same.
* Serious condition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Women suffering from axillary lymphadenectomy due to breast cancer in four spanish hospitals
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
breast cancer-related lymphedema | The agreed date with the participant for the evaluation (second half of 2017)
  Truncated cone formula

SECONDARY OUTCOMES:
functional shoulder limitation | The agreed date with the participant for the evaluation (second half of 2017)
  Shoulder Pain and Disability Index
Symptoms associated with breast cancer-related lymphedema | The agreed date with the participant for the evaluation (second half of 2017)
  Visual Analogic Scale

OTHER OUTCOMES:
Degree of compliance with the prevention program | The agreed date with the participant for the evaluation (second half of 2017)
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Violeta Pajero Otero, MRes, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (5):
- Spain (5):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario Universitario de Cartagena, Cartagena, Murcia
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Castilla-La Mancha University, Toledo

IPD SHARING:
Plan to Share IPD: No